CLINICAL TRIAL: NCT02756663
Title: A Randomized, Triple-arm, Controlled, Open-label, Multicenter Phase II Study Assessing Two Different Doses of Panobinostat in Combination With Carfilzomib and Dexamethasone in Relapsed or Relapsed and Refractory Multiple Myeloma
Brief Title: Panobinostat in Combination With Carfilzomib and Dexamethasone in Relapsed or Relapsed and Refractory Multiple Myeloma
Acronym: PANORAMA-5
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589X2201
Record Dates: First submitted 2016-04-12; First posted 2016-04-29 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; MM; relapsed; relapsed and refractory; panobinostat; LBH589; histone deacetylase inhibitor; carfilzomib; proteasome inhibitor
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Panobinostat; Capsules; carfilzomib; Dexamethasone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: PAN (10mg) + CFZ + Dex (Experimental): Panobinostat (PAN) 10mg orally, combined with carfilzomib (CFZ) 20/56 mg/m2 i.v. and dexamethasone (Dex) 20mg orally, in 4 week cycle
  Interventions: Drug: panobinostat (capsules); Drug: carfilzomib (infusion); Drug: dexamethasone (tablets)
- Arm B: PAN (20mg) + CFZ + Dex (Experimental): Panobinostat (PAN) 20mg orally, combined with carfilzomib (CFZ) 20/56 mg/m2 i.v. and dexamethasone (Dex) 20mg orally, in 4 week cycle
  Interventions: Drug: panobinostat (capsules); Drug: carfilzomib (infusion); Drug: dexamethasone (tablets)
- Arm C: CFZ + Dex (Active Comparator): Carfilzomib (CFZ) 20/56 mg/m2 i.v. and dexamethasone (Dex) 20mg orally, in 4 week cycle
  Interventions: Drug: carfilzomib (infusion); Drug: dexamethasone (tablets)

INTERVENTIONS:
Drug: panobinostat (capsules) — Panobinostat capsules, oral: 10mg, 15mg, 20mg dosing 3x a week, 1 week on / 1 week off, in a 4 week cycle (28 days). Treatment arm A: only capsules of 10mg will be used Treatment arm B: capsules of 10mg and 15mg are foreseen for dose reduction only.
  Other Names: PAN, LBH589
  Arms: Arm A: PAN (10mg) + CFZ + Dex; Arm B: PAN (20mg) + CFZ + Dex
Drug: carfilzomib (infusion) — Carfilzomib infusion; 20 mg/m2 i.v. on C1D1 and C1D2; 56 mg/m2 i.v. on subsequent dosing days (2x a week; 3 weeks on/1 weeks off ); 4 week cycle (28 days)
  Other Names: CFZ
Drug: dexamethasone (tablets) — Dexamethasone tablets p.o. 20 mg on days of carfilzomib infusion (2x week) and on D22 and D23 of each 4 week cycle (28 days)
  Other Names: Dex

SUMMARY:
The purpose of this study is to investigate the anti-myeloma effect of panobinostat given at two different doses (10 mg and 20 mg oral) in combination with carfilzomib (20/56 mg/m2 i.v.) and low dose dexamethasone (20 mg oral) vs carfilzomib plus low-dose dexamethasone in patients with relapsed or relapsed and refractory multiple myeloma. Safety and efficacy will be evaluated. Treatment will be administered in 4-week cycles until patients discontinue due to disease progression or unacceptable toxicity or for other reasons.

Patients who discontinue the study treatment for reasons other than documented disease progression will be followed for disease assessments every 8 weeks until progression. All patients will be followed for survival until 3 years have passed from their entry into the study, or they have discontinued the follow up earlier.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of MM based on IMWG definitions (Rajkumar, 2014)
* Prior treatment with 1 to 3 prior lines of therapy
* Relapsed or relapsed and refractory MM
* Measureable disease at screening based on central laboratory assessment
* ECOG Performance status ≤ 2
* Acceptable lab values prior to starting study treatment

Exclusion Criteria:

* Primary refractory myeloma
* Prior treatment with DAC inhibitors including panobinostat
* Prior treatment with carfilzomib
* Allogeneic stem cell transplant recipient with graft versus host disease (either active or requiring immunosuppression)
* Any concomitant anti-cancer therapy besides the study treatment (bisphosphonates are permitted only if commenced prior to the start of screening period)
* Intolerance to dexamethasone or contraindication to carfilzomib or dexamethasone
* Unresolved diarrhea ≥ CTCAE grade 2 or a medical condition associated with chronic diarrhea (such as irritable bowel syndrome, inflammatory bowel disease)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) using investigator's response assessment | All patients treated for 6 cycles (cycle=28 days)
  The primary endpoint if Overall Response Rate (ORR) using investigator response assessment according to IMWG criteria. The analysis of ORR will be performed after all randomized patients have completed 6 months of study treatment or discontinued treatment earlier.

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) or better as best response using investigator response assessment based on International Myeloma Working Group (IMWG) criteria | All patients treated for 6 cycles (cycle=28 days)
  Investigators' response assessment assessed on IMWG criteria will be used. The VGPR or better rate is defined as the proportion of patients with a confirmed VGPR or better response as their best overall response.
Progression-free survival (PFS) using investigator's response assessment based on IMWG criteria | All patients treated for 6 cycles (cycle=28 days)
  PFS is defined as the time from date of randomization to date of first documented disease progression or death (regardless of cause of death).
Overall survival (OS) | All patients treated for 6 cycles (cycle=28 days)
  OS is defined as the time from date of randomization to the date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last contact.
Time to response (TTR) using investigator's response assessment based on IMWG criteria | All patients treated for 6 cycles (cycle=28 days)
  TTR is the time between date of randomization to the date of first onset of partial response (PR) or better response.
Duration of Response (DOR) using investigator's response assessment based on IMWG criteria | All patients treated for 6 cycles (cycle = 28 days)
  DOR is defined as the duration from the first documented onset of PR or better response the date of first documented disease progression or death due to multiple myeloma. DOR will use only the patients with PR or better as their best response.
Time to progression (TTP) using investigator's response assessment based on IMWG criteria | All patients treated for 6 cycles (cycle = 28 days)
  TTP is defined as the time from the date of randomization to the ate of the first documented disease progression or death due to multiple myeloma.
Time to reach Cmax for panobinostat (PAN) and carfilzomib (CFZ) | All patients treated for 6 cycles (cycle=28 days);
  The maximum (peak) observed plasma concentration after single and multiple dose administration (ng/mL) of PAN and CFZ.
Minimum observed plasma concentration (Cmin) for carfilzomib | All patients treated for 6 cycles (cycle=28 days)
  The minimum (trough) observed plasma concentration after single and multiple dose administration (ng/mL) of PAN and CFZ.
Concentration of panobinostat in blood plasma in 48 hrs after the dose. | All patients treated for 6 cycles (cycle = 28 days)
  The area under the concentration-time curve (AUC) from time zero to 48 hours (ng*h/mL) after the dose of PAN
Total carfilzomib exposure over time in blood plasma . | All patients treated for 6 cycles (cycle=28 days)
  The AUC from time zero to infinity (ng*h/mL) for CFZ.
Health related quality of life (HRQoL) change over time measured by EORTC questionnaire QLQ-C30 and QLQ-MY20 for disease symptoms | All patients treated for 6 cycles (cycle=28 days)
  HRQoL questionnaires are patient reported outcomes, which provide functional assessment of cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals